CLINICAL TRIAL: NCT05391360
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single- and Multiple-dose Study in Healthy Subjects and Chronic Hepatitis B Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics and Antiviral Activity of Freethiadine
Brief Title: Evaluation Freethiadine Tolerance in Healthy Subjects and Patients With Chronic Hepatitis B, Pharmacokinetics Characteristics and Antiviral Activity of Ⅰ Phase of Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HEC160208-HBV-101
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Freethiadine tablets (Experimental): part 1(Health volunteer): single-Dose Study: There will be a total of 5 dose cohorts: 5 mg、10 mg、200 mg(food effect)、400 mg、600 mg; multiple-dose study: 100 mg、200 mg、300 mg、150 mg
  Interventions: Drug: Freethiadine tablets(part I)
- Freethiadine placebo tablets (Placebo Comparator): part 1(Health volunteer): single-Dose Study: There will be a total of 5 dose cohorts: 5 mg、10 mg、200 mg(food effect)、400 mg、600 mg; multiple-dose study: 100 mg、200 mg、300 mg、150 mg
  Interventions: Drug: Freethiadine placebo tablets
- Freethiadine tablet (Experimental): part 2(Patients with chronic hepatitis B): There will be a total of 4 dose cohorts:100 mg、200 mg(BID or QD)、300 mg
  Interventions: Drug: Freethiadine tablets (part II)
- entecavir tablets (Active Comparator): part 2(Patients with chronic hepatitis B): 0.5 mg
  Interventions: Drug: entecavir tablets

INTERVENTIONS:
Drug: Freethiadine tablets(part I) — Subjects will receive either a single dose of Freethiadine on Day 1 only (SAD HV), twice daily dosing of Freethiadine starting on Day 1 through Day 10 (MAD HV)
  Arms: Freethiadine tablets
Drug: Freethiadine tablets (part II) — once or twice daily for consecutive 28 days
  Arms: Freethiadine tablet
Drug: Freethiadine placebo tablets — Subjects will receive either a single dose of Freethiadine on Day 1 only (SAD HV), twice daily dosing of Freethiadine starting on Day 1 through Day 10 (MAD HV)
  Arms: Freethiadine placebo tablets
Drug: entecavir tablets — once daily for consecutive 28 days
  Arms: entecavir tablets

SUMMARY:
The Safety, Tolerability, Pharmacokinetics and antiviral activity Study of Anti hepatitis B virus treatment drug Freethiadine in Healthy subjects and in patients with chronic hepatitis B

ELIGIBILITY:
Inclusion Criteria:

Health volunteer:

1. Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions.
2. subjects and must be 18 to 45 years of age inclusive.
3. Body weight ≥ 45 kg and body mass index（BMI）between 18 and 28 kg / m^2, inclusive.
4. Physical examination and vital signs without clinically significant abnormalities.

Patients with chronic hepatitis B:

1. Sign the informed consent form before the trial and fully understand the contents of the trial, the process and possible adverse reactions.
2. subjects and must be 18 to 65 years of age inclusive.
3. Body mass index（BMI）between 18 and 32 kg / m^2, inclusive.
4. No cirrhosis.

Exclusion Criteria:

Health volunteer:

1. Use of >5 cigarettes per day during the past 3 months.
2. History of alcohol abuse (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits or 100 mL of wine).
3. Donation or loss of blood over 450 mL within 3 months prior to screening.

Patients with chronic hepatitis B:

1. AFP>50 ng/mL.
2. INR>1.5.
3. Positive for Viral hepatitis C, HIV and syphilis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From Days 1-35
  Incidence of adverse events
AUC | Day 1-12
  Maximum plasma concentration of study drugs
HBV DNA | Day 1-35
  Change from baseline in HBV DNA

SECONDARY OUTCOMES:
HBsAg | Day 1-35
  Change from baseline in HBsAg

CONTACTS AND LOCATIONS:
Overall Officials: JinLin Hou, Doctor, Principal Investigator — Southern Hospital of Southern Medical University; JunQI Niu, Doctor, Principal Investigator — The First Hospital of Jilin University; Yanhua Ding, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (2):
- China (2):
  - Southern Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Hospital of Jilin University, Changchun, Jilin